CLINICAL TRIAL: NCT06639620
Title: Effectiveness aNd Use of fosleVOdopa-foscarbidopa in Advanced Parkinson Disease in Real Life Setting
Brief Title: Study To Assess Effectiveness and Adverse Events of Foscarbidopa/ Foslevodopa in Adult Participants With Advanced Parkinson Disease in Real Life Setting
Acronym: ENVOL
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-820
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-08-25 (Actual); Status verified 2025-08

CONDITIONS: Advanced Parkinson Disease
Keywords: Advanced Parkinson disease; Foscarbidopa/ foslevodopa; ABBV-951; LDp/CDp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Foscarbidopa / Foslevodopa: Participants will receive foscarbidopa/ foslevodopa as prescribed by their physician according to local label

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. This study will assess how effective foscarbidopa/ foslevodopa is in treating French adult participants with advanced Parkinson disease under routine clinical practice.

Foslevodopa/foscarbidopa is an approved drug outside of US for the treatment of Parkinson's Disease. Approximately 200 adult participants who are prescribed foslevodopa/foscarbidopa by their doctors will be enrolled across approximately 30 sites in France.

Participants will receive foscarbidopa/ foslevodopa subcutaneous infusion as prescribed by their physician. Participants will be followed for up to 12 months.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with advanced Parkinson disease with motor complications insufficiently controlled by current therapy
* Participants eligible for foscarbidopa / foslevodopa according to French label & regulation.
* Treatment initiation decision prior to and independently from study enrolment

Exclusion Criteria:

* Participants with any contraindication to foscarbidopa / foslevodopa.
* Participants with Mini mental state examination (MMSE) score < 24

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced Parkinson disease treated with Foscarbidopa/ foslevodopa according to label in France
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Parkinson's Disease Questionnaire-8 (PDQ) total score. | Up to approximately 12 months
  Parkinson Disease Questionnaire (PDQ)-8 is an eight-question instrument constructed by taking one question from each domain of PDQ-39: mobility, activities of daily of living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. Each question is scored between 0 and 4 as follows: 0=Never and 4 = Always or cannot do at all. A higher score signifies poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (32):
- France (32):
  - Les Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre /ID# 266843, Strasbourg, Alsace
  - Centre Hospitalier Universitaire Gabriel-Montpied /ID# 267182, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Hôpital La Timone /ID# 265932, Marseille, Bouches-du-Rhone
  - CH de Saint-Brieuc, Paimpol et Tréguier /ID# 266927, Saint-Brieuc, Brittany Region
  - Centre Hospitalier Régional Universitaire de Besançon - Hôpital Jean Minjoz /ID# 266853, Besançon, Doubs
  - CHU Brest /ID# 266405, Brest, Finistere
  - Chu de Limoges /Id# 266043, Limoges, Franche-Comte
  - Hôpitaux Civils de Colmar - Hôpital Pasteur /ID# 266932, Colmar, Grand Est
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Roger Salengro /ID# 265954, Lille, Hauts-de-France
  - Clinique Beausoleil /ID# 266920, Montpellier, Herault
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou /ID# 267665, Rennes, Ille-et-Vilaine
  - CH Bretagne Atlantique /ID# 268308, Vannes, Morbihan
  - Chu De Toulouse - Hopital Pierre Paul Ricquet /ID# 266031, Toulouse, Occitanie
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 266034, Créteil, Paris
  - Centre Hospitalier d'Avignon /ID# 266369, Avignon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Côte Basque /ID# 266846, Bayonne, Pyrenees-Atlantiques
  - les Hospices Civils de Lyon (HCL) /ID# 266404, Lyon, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 266039, Amiens, Somme
  - Centre Hospitalier Intercommunal Toulon /ID# 266397, Toulon, Var
  - Centre Hospitalier Emile Durkheim - Site Plateau de la Justice /ID# 267183, Épinal, Vosges
  - Cabinet de Neurologie /ID# 268309, Versailles, Yvelines
  - Ch Bethune - Beuvry /Id# 265994, Béthune
  - Centre hospitalier de Brive /ID# 265952, Brive-la-Gaillarde
  - Centre Hospitalier Public du Cotentin - Hôpital Pasteur /ID# 265950, Cherbourg
  - CH Haguenau /ID# 266029, Haguenau
  - CHRU de NANCY /ID# 266385, Nancy
  - Centre Hospitalier Universitaire de Nîmes - Hôpital Universitaire Carémeau /ID# 266375, Nîmes
  - Hôpital Fondation Adolphe de Rothschild /ID# 266373, Paris
  - CHU de Rouen /ID# 266390, Rouen
  - CHU de Nantes - Hopital Nord Laennec /ID# 266036, Saint-Herblain
  - Centre Hospitalier de Saint Malo /ID# 265948, St-Malo
  - Centre Hospitalier de Valenciennes /ID# 266400, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-820